CLINICAL TRIAL: NCT04362813
Title: Phase 3 Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of Canakinumab on Cytokine Release Syndrome in Patients With COVID-19-induced Pneumonia (CAN-COVID)
Brief Title: Study of Efficacy and Safety of Canakinumab Treatment for CRS in Participants With COVID-19-induced Pneumonia
Acronym: CAN-COVID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CACZ885D2310; 2020-001370-30 (EudraCT Number)
Record Dates: First submitted 2020-04-24; First posted 2020-04-27 (Actual); Results first posted 2021-08-16 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Cytokine Release Syndrome (CRS) in Patients With COVID-19-induced Pneumonia
Keywords: COVID-19; cytokine release syndrome; SARS-CoV-2; canakinumab; COVID; coronavirus; CAN-COVID; pneumonia; CRS
MeSH Terms: conditions — Cytokine Release Syndrome; COVID-19; Coronavirus Infections; Pneumonia | interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Canakinumab (Experimental): Canakinumab 450 mg for body weight 40-<60 kg, 600 mg for 60-80 kg or 750 mg for >80 kg in 250 mL of 5% dextrose infused IV over 2 hours. Single dose on Day 1.
  Interventions: Drug: Canakinumab
- Placebo (Placebo Comparator): 250 mL of 5% dextrose infused IV over 2 hours. Single dose on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canakinumab — Canakinumab 450 mg for body weight 40-<60 kg, 600 mg for 60-80 kg or 750 mg for >80 kg in 250 mL of 5% dextrose infused IV over 2 hours. Single dose on Day 1.
  Other Names: ACZ885
  Arms: Canakinumab
Drug: Placebo — 250 mL of 5% dextrose infused IV over 2 hours. Single dose on Day 1.
  Arms: Placebo

SUMMARY:
This was a multicenter, randomized, double-blind, placebo-controlled study to assess the efficacy and safety of canakinumab plus standard-of-care (SOC) compared with placebo plus SOC in patients with COVID-19-induced pneumonia and cytokine release syndrome (CRS).

DETAILED DESCRIPTION:
This was a Phase III, multicenter, randomized, double-blind, placebo-controlled study to assess the efficacy and safety of canakinumab in patients with COVID-19-induced pneumonia and cytokine release syndrome (CRS). The study enrolled patients to canakinumab or placebo, in addition to standard of care (SOC) per local practice, which may have included anti-viral treatment, corticosteroids and/or supportive care.

Patients who met the inclusion/exclusion criteria were randomized in a 1:1 ratio to either canakinumab + SOC or placebo + SOC and were dosed immediately after ensuring that the patient met all eligibility criteria. Patients in the canakinumab arm were dosed on Day 1 with canakinumab 450 mg for body weight of 40-<60 kg, 600 mg for 60-80 kg or 750 mg for >80 kg in 250 mL of 5% dextrose infused IV over 2 hours. Patients in the placebo arm were administered with 250 mL of 5% dextrose infused IV over 2 hours.

The study included:

* Screening period of 0-1 day
* Study period from initial dose on Day 1 to Day 29 or hospital discharge
* Follow-up to Day 127 The primary objective was to demonstrate the benefit of canakinumab + SOC in increasing the chance of survival without ever requiring invasive mechanical ventilation among patients with COVID-19-induced pneumonia and CRS.

ELIGIBILITY:
Key inclusion Criteria:

* Adults ≥ 18 years old (for US only: patients ≥ 12 years old, although no children ever enrolled. This was an adult trial.)
* Body weight ≥40 kg
* Informed consent must be obtained prior to participation in this study. For US patients 12 - < 18 years old; parent/guardian consent must be obtained and assent if applicable.
* Clinically diagnosed with SARS-CoV-2 virus by PCR or by other approved diagnostic methodology
* Hospitalized with COVID-19-induced pneumonia evidenced by chest x-ray or CT scan with pulmonary infiltrates
* SpO2 ≤ 93% on room air or arterial oxygen partial pressure (PaO2)/ fraction of inspired oxygen (FiO2) < 300mmHg
* C-reactive protein ≥20 mg/L or ferritin level ≥600 µg/L

Key exclusion Criteria:

* History of hypersensitivity to canakinumab or to biologic drugs
* Intubated and on mechanical ventilation (invasive) at time of randomization
* Treatment with immunomodulators or immunosuppressant drugs, including but not limited to tocilizumab, TNF inhibitors and anti-IL-17 agents within 5 half-lives or 30 days (whichever is longer) prior to randomization with the exception of anakinra which is excluded within 5 half-lives only. Note: Immunomodulators (topical or inhaled) for asthma and atopic dermatitis and corticosteroids (any route of administration) are permitted.
* Suspected or known untreated active bacterial, fungal, viral, or parasitic infection with the exception of COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartiis Pharmaceuticals
Locations (30):
- United States (13):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Glendale, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Brooklyn, New York
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Tacoma, Washington
- Novartis Investigative Site, Toulouse, France
- Italy (2):
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Cona, FE
- Russia (6):
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, S-Petersburg
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Sestroretsk
- Spain (4):
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, San Sebastián de los Reyes, Madrid
  - Novartis Investigative Site, Madrid
- United Kingdom (4):
  - Novartis Investigative Site, Barnet
  - Novartis Investigative Site, Coventry
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Sedhai YR, Sears M, Vecchie A, Bonaventura A, Greer J, Spence K, Tackett H, Turner J, Pak M, Patel N, Black M, Wohlford G, Clary RE, Duke C, Hardin M, Kemp H, Priday A, Sims EK Jr, Mihalick V, Ho AC, Ibe I, Harmon M, Markley R, Van Tassell B, Abbate A. Clinical trial enrollment at a rural satellite hospital during COVID-19 pandemic. J Clin Transl Sci. 2021 Apr 8;5(1):e136. doi: 10.1017/cts.2021.777. eCollection 2021. PMID 34367680
- [Derived] Caricchio R, Abbate A, Gordeev I, Meng J, Hsue PY, Neogi T, Arduino R, Fomina D, Bogdanov R, Stepanenko T, Ruiz-Seco P, Gonzalez-Garcia A, Chen Y, Li Y, Whelan S, Noviello S; CAN-COVID Investigators. Effect of Canakinumab vs Placebo on Survival Without Invasive Mechanical Ventilation in Patients Hospitalized With Severe COVID-19: A Randomized Clinical Trial. JAMA. 2021 Jul 20;326(3):230-239. doi: 10.1001/jama.2021.9508. PMID 34283183
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=971

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part at 39 investigative sites in 6 countries.
  While patient flow shows 454 participants enrolled, only 451 randomized. 3 were "mis-randomized" i.e. assigned a randomization number in error and not treated.
Pre-assignment Details: Participants were screened within 24 hours prior to enrollment.
Period: Overall Study
Arm/Group | Canakinumab | Placebo
Started (Ranomized participants) | 227 | 227
Safety Set (The Safety Set included all participants who received at least one dose of double-blind treatment) | 225 | 223
Completed Day 29 | 211 | 206
Completed | 209 | 202
Not Completed | 18 | 25
Not completed — Death | 12 | 16
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Protocol Violation | 0 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Enrolled but did not receive treatment | 2 | 4

BASELINE CHARACTERISTICS:
Population: While patient flow and baseline measure tables show 454 participants enrolled, only 451 randomized. 3 were "mis-randomized" i.e. assigned a randomization number in error and not treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Canakinumab | Placebo | Total
Number analyzed (Participants) | 227 | 227 | 454
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (14.55) | 57.8 (13.89) | 58.2 (14.21)
Age, Customized [Count of Participants; unit: Participants]
  < 18 years | 0 | 0 | 0
  Between 18 and 64 years | 149 | 155 | 304
  >=65 years | 78 | 72 | 150
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 95 | 187
  Male | 135 | 132 | 267
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 8 | 11
  Asian | 10 | 9 | 19
  Native Hawaiian or Other Pacific Islander | 1 | 5 | 6
  Black or African American | 35 | 37 | 72
  White | 159 | 156 | 315
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 19 | 12 | 31

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Survived Without Requiring Invasive Mechanical Ventilation From Day 3 to Day 29, Primary Analysis
Description: Number of responders who survived without requiring invasive mechanical ventilation from Day 3 to Day 29. An early dropout without requiring invasive mechanical ventilation is considered as a responder if discharged from hospital with 9-point ordinal scale<=1 or with last 9-point ordinal scale on/after Day 15 better than baseline.
Time Frame: Day 3 to Day 29
Population: Randomized participants with at least one assessment of the 9-point ordinal scale between Day 3 and Day 29 (where value 0 = uninfected, and 8 = death)
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 223 | 223
Participants | 198 | 191
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; Odds ratio is based on a Logistic regression model adjusted by treatment, region (North America vs Europe), and baseline 9-point ordinal scale (<=4, >=5); Test type: Superiority; p = 0.2874, Regression, Logistic; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.76 to 2.54]

2. Secondary Outcome: COVID-19-related Death After Study Treatment
Description: Participants with COVID-19 related (as assessed by investigator) death up to Day 29
Time Frame: 29 days
Population: All randomized participants including those who did not receive any dose, as per intent-to-treat principle, and excluding early dropouts if the last available 9-point ordinal scale >1 (including non-COVID-19 related death)
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 223 | 222
Participants | 11 | 16
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.3303, Regression, Logistic; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.30 to 1.50]

3. Secondary Outcome: Geometric Mean Ratio to Baseline in the C-reactive Protein (CRP)
Description: Measurement of C Reactive Protein (mg/L), Serum Or Plasma over time. The level of C-reactive protein (CRP), which can be measured in the blood, increases when there's inflammation in the body. Lower values of ratio to baseline in the CRP indicates less inflammation. The ratio to baseline at each time point (day) for each patient is calculated as the level of a specific biomarker at the time point divided by the baseline level of the biomarker, where baseline is the last non-missing value before study treatment. The geometric mean of ratio to baseline at each time point for each treatment group is calculated by first averaging the logarithms of the ratios to baseline and then take the exponential function of the same base.
Time Frame: Over time and up to day 29: Baseline, Day 2, Day 3, Day 5, Day 7, Day 9, Day 11, Day 13, Day 15, Day 17, Day 19, Day 21, Day 23, Day 25, Day 27 and Day 29.
Population: Randomized participants with a valid assessment for the outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 227 | 227
ratio
  Day 2: number analyzed (Participants) | 219 | 214
  Day 2 | 0.726 [0.671 to 0.786] | 0.785 [0.722 to 0.853]
  Day 3: number analyzed (Participants) | 208 | 194
  Day 3 | 0.479 [0.430 to 0.534] | 0.649 [0.578 to 0.729]
  Day 5: number analyzed (Participants) | 197 | 193
  Day 5 | 0.255 [0.222 to 0.292] | 0.384 [0.325 to 0.454]
  Day 7: number analyzed (Participants) | 168 | 179
  Day 7 | 0.160 [0.129 to 0.198] | 0.238 [0.195 to 0.290]
  Day 9: number analyzed (Participants) | 132 | 141
  Day 9 | 0.131 [0.101 to 0.171] | 0.159 [0.126 to 0.201]
  Day 11: number analyzed (Participants) | 112 | 111
  Day 11 | 0.099 [0.073 to 0.133] | 0.133 [0.096 to 0.185]
  Day 13: number analyzed (Participants) | 86 | 86
  Day 13 | 0.108 [0.072 to 0.162] | 0.141 [0.087 to 0.228]
  Day 15: number analyzed (Participants) | 74 | 72
  Day 15 | 0.133 [0.086 to 0.205] | 0.149 [0.088 to 0.252]
  Day 17: number analyzed (Participants) | 47 | 50
  Day 17 | 0.123 [0.069 to 0.220] | 0.289 [0.189 to 0.441]
  Day 19: number analyzed (Participants) | 30 | 33
  Day 19 | 0.123 [0.059 to 0.255] | 0.368 [0.227 to 0.598]
  Day 21: number analyzed (Participants) | 17 | 20
  Day 21 | 0.115 [0.053 to 0.247] | 0.296 [0.164 to 0.533]
  Day 23: number analyzed (Participants) | 26 | 28
  Day 23 | 0.106 [0.036 to 0.311] | 0.400 [0.201 to 0.796]
  Day 25: number analyzed (Participants) | 11 | 17
  Day 25 | 0.126 [0.024 to 0.633] | 0.368 [0.160 to 0.846]
  Day 27: number analyzed (Participants) | 11 | 14
  Day 27 | 0.175 [0.041 to 0.743] | 0.331 [0.152 to 0.720]
  Day 29: number analyzed (Participants) | 11 | 14
  Day 29 | 0.240 [0.052 to 1.106] | 0.258 [0.121 to 0.551]

4. Secondary Outcome: Geometric Mean Ratio to Baseline in the D-dimer
Description: Clinical chemistry measurement D-Dimer (mg/L FEU), Blood in a blood sample over time
  D-dimer is one of the protein fragments produced when a blood clot gets dissolved in the body. The ratio to baseline at each time point (day) for each patient is calculated as the level of a specific biomarker at the time point divided by the baseline level of the biomarker, where baseline is the last non-missing value before study treatment. The geometric mean of ratio to baseline at each time point for each treatment group is calculated by first averaging the logarithms of the ratios to baseline and then take the exponential function of the same base.
Time Frame: as for outcome 3
Population: FAS
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 227 | 227
ratio
  Day 2: number analyzed (Participants) | 197 | 190
  Day 2 | 1.032 [0.910 to 1.170] | 1.028 [0.948 to 1.114]
  Day 3: number analyzed (Participants) | 192 | 172
  Day 3 | 0.992 [0.866 to 1.135] | 1.188 [1.004 to 1.242]
  Day 5: number analyzed (Participants) | 172 | 169
  Day 5 | 1.094 [0.971 to 1.233] | 1.188 [1.061 to 1.330]
  Day 7: number analyzed (Participants) | 144 | 160
  Day 7 | 1.038 [0.851 to 1.267] | 1.244 [1.088 to 1.422]
  Day 9: number analyzed (Participants) | 120 | 129
  Day 9 | 1.164 [0.961 to 1.410] | 1.184 [1.003 to 1.422]
  Day 11: number analyzed (Participants) | 97 | 95
  Day 11 | 1.162 [0.929 to 1.453] | 1.115 [0.896 to 1.388]
  Day 13: number analyzed (Participants) | 73 | 76
  Day 13 | 1.135 [0.891 to 1.447] | 1.184 [0.927 to 1.513]
  Day 15: number analyzed (Participants) | 61 | 68
  Day 15 | 1.100 [0.800 to 1.514] | 1.078 [0.862 to 1.349]
  Day 17: number analyzed (Participants) | 39 | 47
  Day 17 | 1.033 [0.698 to 1.528] | 1.384 [1.041 to 1.838]
  Day 19: number analyzed (Participants) | 24 | 28
  Day 19 | 1.520 [0.853 to 2.711] | 1.446 [1.005 to 2.081]
  Day 21: number analyzed (Participants) | 21 | 24
  Day 21 | 1.431 [0.770 to 2.659] | 1.443 [0.958 to 2.172]
  Day 23: number analyzed (Participants) | 14 | 18
  Day 23 | 1.208 [0.495 to 2.950] | 1.521 [1.093 to 2.118]
  Day 25: number analyzed (Participants) | 9 | 14
  Day 25 | 2.670 [0.362 to 3.891] | 1.808 [0.969 to 3.371]
  Day 27: number analyzed (Participants) | 9 | 12
  Day 27 | 1.785 [0.644 to 4.949] | 2.262 [1.008 to 5.075]
  Day 29: number analyzed (Participants) | 9 | 12
  Day 29 | 1.818 [0.627 to 5.270] | 2.441 [0.912 to 6.534]

5. Secondary Outcome: Geometric Mean Ratio to Baseline in Ferritin
Description: Clinical chemistry measurement for amount of ferritin (ug/L) in Serum. The ratio to baseline at each time point (day) for each patient is calculated as the level of a specific biomarker at the time point divided by the baseline level of the biomarker, where baseline is the last non-missing value before study treatment. The geometric mean of ratio to baseline at each time point for each treatment group is calculated by first averaging the logarithms of the ratios to baseline and then take the exponential function of the same base.
Time Frame: as for outcome 3
Population: Randomized participants with a valid assessment for the outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 227 | 227
ratio
  Day 2: number analyzed (Participants) | 202 | 198
  Day 2 | 0.996 [0.953 to 1.040] | 1.014 [0.972 to 1.058]
  Day 3: number analyzed (Participants) | 185 | 177
  Day 3 | 0.921 [0.870 to 0.976] | 1.014 [0.954 to 1.077]
  Day 5: number analyzed (Participants) | 171 | 177
  Day 5 | 0.825 [0.765 to 0.889] | 0.879 [0.810 to 0.953]
  Day 7: number analyzed (Participants) | 153 | 163
  Day 7 | 0.761 [0.701 to 0.826] | 0.815 [0.742 to 0.896]
  Day 9: number analyzed (Participants) | 119 | 128
  Day 9 | 0.676 [0.609 to 0.751] | 0.764 [0.679 to 0.859]
  Day 11: number analyzed (Participants) | 98 | 97
  Day 11 | 0.618 [0.548 to 0.698] | 0.735 [0.637 to 0.849]
  Day 13: number analyzed (Participants) | 81 | 72
  Day 13 | 0.582 [0.501 to 0.675] | 0.684 [0.563 to 0.830]
  Day 15: number analyzed (Participants) | 67 | 65
  Day 15 | 0.535 [0.448 to 0.638] | 0.618 [0.510 to 0.750]
  Day 17: number analyzed (Participants) | 43 | 45
  Day 17 | 0.534 [0.449 to 0.634] | 0.641 [0.495 to 0.832]
  Day 19: number analyzed (Participants) | 30 | 29
  Day 19 | 0.545 [0.420 to 0.707] | 0.644 [0.464 to 0.893]
  Day 21: number analyzed (Participants) | 24 | 24
  Day 21 | 0.514 [0.377 to 0.700] | 0.644 [0.439 to 0.944]
  Day 23: number analyzed (Participants) | 15 | 19
  Day 23 | 0.469 [0.294 to 0.749] | 0.692 [0.432 to 1.109]
  Day 25: number analyzed (Participants) | 9 | 16
  Day 25 | 0.542 [0.310 to 0.945] | 0.745 [0.524 to 1.059]
  Day 27: number analyzed (Participants) | 10 | 13
  Day 27 | 0.490 [0.299 to 0.802] | 0.809 [0.480 to 1.363]
  Day 29: number analyzed (Participants) | 9 | 16
  Day 29 | 0.543 [0.212 to 1.393] | 0.517 [0.298 to 0.896]

6. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Number of participants with treatment emergent adverse events, including changes from baseline in vital signs and laboratory results qualifying and reported as adverse events.
  Safety was monitored from the canakinumab or placebo dose (Day 1) up to 126 days post-dose (Day 127).
Time Frame: Up to day 127
Population: Safety Set comprises all participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 225 | 223
Participants | 141 | 140

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study at day 127
Description: Adverse Events (AEs) are any untoward sign or symptom that occurs during the study treatment. Adverse events and all-cause mortality are evaluated in the Safety Set that includes all participants who received at least one dose of double-blind treatment.
Arm/Group | Canakinumab | Placebo
All-Cause Mortality (participants affected / at risk) | 22/225 | 26/223
Serious Adverse Events (participants affected / at risk) | 47/225 | 53/223
Other Adverse Events (participants affected / at risk) | 15/225 | 19/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (N=225) | Placebo (N=223)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 2
Coagulopathy (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 2
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 1
Cardiopulmonary failure (Cardiac disorders) | 2 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Pulseless electrical activity (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal motility disorder (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Antibiotic associated colitis (Infections and infestations) | 2 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 3
COVID-19 pneumonia (Infections and infestations) | 1 | 3
Candida infection (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 1 | 0
Enterocolitis viral (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 3
Pneumonia bacterial (Infections and infestations) | 1 | 2
Pneumonia escherichia (Infections and infestations) | 0 | 1
Pneumonia fungal (Infections and infestations) | 1 | 0
Pneumonia haemophilus (Infections and infestations) | 0 | 1
Pneumonia pseudomonal (Infections and infestations) | 0 | 2
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 3 | 2
Septic shock (Infections and infestations) | 3 | 5
Staphylococcal bacteraemia (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1
Wound necrosis (Injury, poisoning and procedural complications) | 1 | 0
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Bipolar disorder (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 7
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Renal injury (Renal and urinary disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 12 | 13
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 1
Haemodynamic instability (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 3
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (N=225) | Placebo (N=223)
Anaemia (Blood and lymphatic system disorders) | 6 | 12
Hypotension (Vascular disorders) | 12 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Publications from a single-site are postponed until publication of the pooled clinical trial data (i.e., data from all sites) or disclosure of trial results in their entirety

DOCUMENTS (2):
  • Study Protocol (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT04362813/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/13/NCT04362813/SAP_001.pdf